CLINICAL TRIAL: NCT00064272
Title: Phase II Trial Of Encapsulized Ginger As A Treatment For Chemotherapy-Induced Nausea and Vomiting AKA IRB 2003-213
Brief Title: UMCCOP 02-01 Ginger in Treating Nausea and Vomiting in Patients Receiving Chemotherapy for Cancer
Acronym: IRB 2003-551
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000310163; P30CA046592 (NIH); CCUM-0201
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

ARMS (3):
- Arm I (Experimental): Patients receive lower-dose oral ginger twice daily.
  Interventions: Drug: ginger extract
- Arm II (Experimental): Patients receive higher-dose oral ginger twice daily.
  Interventions: Drug: ginger extract
- Arm III (Placebo Comparator): Patients receive oral placebo twice daily.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ginger extract — Given orally
  Arms: Arm I; Arm II
Other: placebo — Given orally
  Arms: Arm III

SUMMARY:
RATIONALE: The herb ginger may help to reduce or prevent nausea and vomiting in patients receiving chemotherapy for cancer.

PURPOSE: This randomized phase II trial is studying how well ginger works in reducing or preventing nausea and vomiting in patients who are receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the prevalence and severity of delayed nausea and vomiting in patients with cancer undergoing chemotherapy treated with lower-dose ginger vs higher-dose ginger vs placebo.

Secondary

* Compare the prevalence and severity of acute nausea and vomiting in patients treated with these regimens.
* Compare the safety of these regimens in these patients.
* Determine whether patients can determine if they are receiving placebo or study drug, and by which variable (e.g., taste, smell, or decrease in nausea and vomiting).

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 3 treatment arms. Patients are stratified according to concurrent antiemetic type (5-HT_3 antagonist vs NK1 antagonist).

* Arm I: Patients receive lower-dose oral ginger twice daily.
* Arm II: Patients receive higher-dose oral ginger twice daily.
* Arm III: Patients receive oral placebo twice daily. In all arms, treatment begins immediately after the chemotherapy treatment and continues for 3 days.

Patients are followed at 1 week.

PROJECTED ACCRUAL: A total of 180 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of cancer
* Currently receiving chemotherapy* containing any chemotherapeutic agent at any dose and experiencing nausea and/or vomiting of any severity (delayed or acute)

  * Chemotherapy regimens may be given orally, IV, or by continuous infusion (single day regimens only)
* Must have received at least 1 prior chemotherapy* course containing any chemotherapeutic agent and meets the following criteria:

  * Agent is the same that is scheduled for the next round of chemotherapy
  * Experienced nausea and/or vomiting of any severity (delayed or acute)
* Must be planning to receive a concurrent 5-HT_3 receptor antagonist antiemetic (e.g., ondansetron, granisetron, dolasetron mesylate, or palanosetron) or antiemetic aprepritant (e.g., Emend®) while on chemotherapy
* No symptomatic brain metastases NOTE: *Chemotherapy may be adjuvant, neoadjuvant, curative, or palliative

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No history of bleeding disorder
* No thrombocytopenia

Hepatic

* Not specified

Renal

* Not specified

Gastrointestinal

* Able to swallow capsules
* No gastric ulcer
* No clinical evidence of current or impending bowel obstruction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to understand English
* Able to complete study questionnaires
* No allergy to ginger

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy regimens with multiple day doses

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy that is classified as high or intermediate risk of causing vomiting, including radiotherapy to any of the following areas:

  * Total body irradiation
  * Hemi-body
  * Upper abdomen
  * Abdominal-pelvic mantle
  * Cranium (radiosurgery)
  * Craniospinal radiotherapy

Surgery

* Not specified

Other

* More than 1 week since prior ginger (teas, capsules, tinctures)
* No other concurrent ginger (teas, capsules, tinctures)

  * Concurrent foods made with small amounts (no more than ¼ teaspoon) of ginger (powdered or fresh) allowed
* No concurrent therapeutic-doses of warfarin, aspirin, or heparin

  * Concurrent low-dose warfarin to maintain peripheral or central venous access, low-dose aspirin (≤ 81 mg), or low-dose heparin allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Most efficacious dose
Safety
Ability to distinguish between receiving placebo or study drug and variables involved (e.g., taste, smell, or decrease in nausea and vomiting)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna Zick, MPH, ND, Study Chair — University of Michigan Rogel Cancer Center
Locations (6):
- United States (5):
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - University of Michigan Cancer Center CCOP Research Base, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - MBCCOP - Our Lady of Mercy Cancer Center, The Bronx, New York
- MBCCOP - San Juan, San Juan, Puerto Rico